CLINICAL TRIAL: NCT03746847
Title: Somatostatin Receptor Imaging in Patients With Suspected Cardiac Sarcoidosis
Brief Title: PET Imaging in Patients With Suspected Cardiac Sarcoidosis
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Advanced Accelerator Applications (Industry)
Responsible Party: Principal Investigator, Paco Bravo, MD, Assistant Professor of Radiology at the Hospital of the University of Pennsylvania, University of Pennsylvania
Other Study IDs: 829715
Record Dates: First submitted 2018-10-29; First posted 2018-11-20 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Cardiac Sarcoidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Suspected Cardiac Sarcoidosis: patients with biopsy proven or suspected sarcoidosis (based on standard clinical imaging findings).
  Interventions: Drug: Gallium-68 DOTATATE

INTERVENTIONS:
Drug: Gallium-68 DOTATATE — Gallium-68 DOTATATE is a radioactive tracer, a type of imaging drug that is labeled with a radioactive tag and injected into the body, which is approved by the U.S. Food and Drug Administration (FDA) to diagnose certain tumors.

SUMMARY:
Gallium-68 DOTATATE is a radioactive tracer, a type of imaging drug that is labeled with a radioactive tag and injected into the body, which is approved by the U.S. Food and Drug Administration (FDA) to diagnose certain tumors. The study will see how the tracer is taken up in your heart before and after treatment using an imaging scan called Positron Emission Tomography / Computed Tomography (PET/CT). Investigators are doing this research study to find out if DOTATATE can help doctors diagnose people with cardiac (heart) sarcoidosis better as well as serve as a follow-up monitoring tool for a response to therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be ≥ 18 years of age
2. History of biopsy-proven sarcoidosis OR suspected sarcoidosis based on standard clinical imaging (e.g. FDG PET/CT, MRI) without biopsy confirmation
3. Clinical suspicion of cardiac involvement defined as the presence of any of the following:

   1. High degree A-V nodal block
   2. Complete bundle branch block
   3. Reduced left or right ventricular systolic fusion
   4. Any cardiac arrhythmia
   5. Chest pain, dyspnea or syncope without clear etiology
4. FDG PET/CT scan demonstrating abnormal myocardial FDG uptake
5. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures

Exclusion Criteria:

1. Females who are pregnant or breast feeding at the time of screening will not be eligible for this study; a urine pregnancy test will be performed in women of child-bearing potential at screening.
2. History of neuroendocrine tumors
3. Currently taking the medication Octreotide
4. Currently on total parenteral nutrition (TPN)
5. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
6. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Suspected Cardiac Sarcoidosis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Dotatate SUVmax activity in the heart | 3 years
  The standardized uptake value (SUV) is a nuclear medicine unit commonly used to distinguish between "normal" and "abnormal" levels of tissue uptake.

SECONDARY OUTCOMES:
Change in Dotatate SUVmax activity in the heart on follow-up PET/CT scan compared to baseline | 3 years
  Dotatate activity (in SUVmax units) in the heart will be measured at baseline and then again at least 3 months after immunotherapy initiation in subjects with suspected cardiac sarcoidosis

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided